CLINICAL TRIAL: NCT06859970
Title: An Early Feasibility Study Evaluation of an Implant Free Interatrial Shunt to Improve Heart Failure
Acronym: EASE HF2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InterShunt Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-00007
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Failure NYHA Class III; Heart Failure With Reduced Ejection Fraction; Ambulatory Heart Failure, NYHA Class IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PAS-C System (Experimental): The PAS-C System is a catheter designed to remove a small section of septal tissue in the interatrial septum to treat heart failure patients without the need for a permanent implant.
  Interventions: Device: PAS-C System

INTERVENTIONS:
Device: PAS-C System — All patients will undergo catheterization with the PAS-C System to create an interatrial shunt to reduce left atrial pressure in the heart.

SUMMARY:
The purpose of this early feasibility study is to evaluate the safety and feasibility of the device for percutaneous shunting of the interatrial septum and improvement of heart failure related symptoms. The primary goal is to determine if the device is safe to use. The findings from this study may be used to refine the intended patient population, the design of the device, or develop a subsequent randomized study.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm early feasibility study (EFS) to evaluate the safety of the InterShunt PAS-C System in subjects with heart failure, and the feasibility of PAS-C to improve heart failure related symptoms. The device is used to create an interatrial shunt by removing septal tissue to reduce left atrial pressure. There is no permanent implant. Enrollment will include 20 subjects with documented heart failure who may benefit from the reduction of left atrial pressure. The primary objective of this study is to characterize the safety of using the PAS-C System by evaluating the proportion of subjects who experience a major adverse cardiac or cerebrovascular event or systemic embolization through one month after the procedure. The findings from this study will be used to develop a subsequent pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* NYHA Class II at screening with a prior history of greater than NYHA Class II, OR NYHA Class III at screening, OR ambulatory Class IV at screening: with documented medical history of heart failure for at least 6 months prior to the screening visit.
* At least one hospitalization for heart failure OR treatment with IV diuretics for heart failure OR elevated BNP in the prior 12 months.
* Receiving maximally tolerated guideline directed medical therapy for Heart Failure management.
* LVEF ≥ 20% and ≤ 40% according to baseline echocardiography.
* Resting right heart catheterization demonstrates elevated PCWP compared to right atrial pressure.

Exclusion Criteria:

* Any of the following within the prior 6 months: Stroke, thromboembolism, severe or advanced heart failure such as Stage D heart failure, non-ambulatory NYHA Class IV, cardiac index less than 1.8 L/min/m2, LVEDD > 8 cm, or received inotropic therapy for LVEF less than 20%.
* Any of the following within the prior 3 months: Myocardial infarction percutaneous cardiac intervention, CABG, on cardiac transplant list, cardiac resynchronization therapy implant, AICD implant, or indicated for coronary revascularization at the time of enrollment.
* Transseptal procedure or percutaneous cardiac intervention planned within the next 6 months.
* Chronic pulmonary disease requiring continuous home oxygen or hospitalization within the prior 12 months for pulmonary disease.
* Patent foramen ovale (PFO) device or atrial septal defect (ASD) device.
* BMI > 40.
* Anatomic anomaly that precludes creation of interatrial shunt.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Measure of major safety events in the periprocedural timeframe | Through one month post procedure
  Proportion of subjects who experience a major adverse cardiac or cerebrovascular event or systemic embolization

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - St. Bernard's Healthcare, Jonesboro, Arkansas
  - Los Robles Health System, Thousand Oaks, California
  - Ascension St. Vincent Hospital, Indianapolis, Indiana
  - Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Methodist Healthcare, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No